CLINICAL TRIAL: NCT02983201
Title: A Clinical Study of Acupuncture Comprehensive Therapy on Common Orthopedic Pain Syndromes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW13-348
Record Dates: First submitted 2016-10-06; First posted 2016-12-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Pain
Keywords: Orthopedic Pain Syndromes; Thumbtack Intra-dermal Needle; Filiform needle; Acupuncture
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- filiform needle (Active Comparator): Patients will receive filiform needle treatment only.During the study period, a maximum of two courses of acupuncture therapy, consisting of 7 sessions each, will be administered. Treatment will be given twice per week. After completing the first course of 7 sessions, there will be a break of one week, at the end of which the second course will commence. Treatment will come to a halt as soon as the pain has totally subsided.
  Interventions: Other: filiform needle
- thumbtack needle+filiform needle (Experimental): Thumbtack intra-dermal needle will be applied to selected acupuncture points after filiform needle treatment. The thumbtack needle will remain embedded in the patient's dermal part for 2-3 days as per instruction.During the study period, a maximum of two courses of acupuncture therapy, consisting of 7 sessions each, will be administered. Treatment will be given twice per week. After completing the first course of 7 sessions, there will be a break of one week, at the end of which the second course will commence. Treatment will come to a halt as soon as the pain has totally subsided.
  Interventions: Other: filiform needle; Other: thumbtack needle

INTERVENTIONS:
Other: filiform needle — Patients will receive filiform needle treatment only.During the study period, a maximum of two courses of acupuncture therapy, consisting of 7 sessions each, will be administered. Treatment will be given twice per week. After completing the first course of 7 sessions, there will be a break of one week, at the end of which the second course will commence. Treatment will come to a halt as soon as the pain has totally subsided.
Other: thumbtack needle — Thumbtack intra-dermal needle will be applied to selected acupuncture points after filiform needle treatment. The thumbtack needle will remain embedded in the patient's dermal part for 2-3 days as per instruction.During the study period, a maximum of two courses of acupuncture therapy, consisting of 7 sessions each, will be administered. Treatment will be given twice per week. After completing the first course of 7 sessions, there will be a break of one week, at the end of which the second course will commence. Treatment will come to a halt as soon as the pain has totally subsided.
  Arms: thumbtack needle+filiform needle

SUMMARY:
The objective of this trial is to further confirm and assess the efficacy of filiform needle therapy on the common orthopedic pain syndromes and investigate whether or not thumbtack needle therapy could further enhance the clinical efficacy and pain healing effect of the filiform needle therapy.

DETAILED DESCRIPTION:
Thumbtack Intra-dermal Needle is a type of intra-dermal needle with a round thumbtack like needle head that is perpendicular to the needle and its sharp end. It is also named as Push-pin Intra-dermal Needle. The Thumbtack Intra-dermal Needle is designed to be embedded in the dermal part of the patients'body for a prolong period to provide continuous stimulation, it is a further development of the treatment method of retaining the filiform needle in the patients'body. The main purpose of embedding the needle in the patients' body for a prolong period of time is to enhance the effect of acupuncture, and improve its clinical efficacy. After the Thumbtack Intra-dermal Needle is applied to the acupuncture point, the needle will be fastened by adhesive tape on the skin surface, and embedded in the dermal part of the patient's body for a period of time. Currently, Thumbtack Intra-dermal Needle is widely used in clinical application. On April 23, 2008, the State Administration of Quality Supervision, Inspection and Quarantine of the People's Republic of China, together with the China National Standardization Management Committee, released the GB standard of applying Intra-dermal Needle: The national standard of the People's Republic of China - Acupuncture and Practices, Part 8: Intra-dermal Needle (GB/T 21709. 8-2008).

Filiform needle is the most common needle used for acupuncture, and it is commonly accepted as the primary tool to perform acupuncture. Traditional Acupuncture (using filiform needle)is proven to be effective in pain management. In 2003, World Health Organization(WHO) confirmed that "There is significant neurophysiological evidence that supports the the notion that acupuncture is capable of modulating pain sensation". Relatively fewer research and study has been done on efficacy of Intra-dermal needle in pain management.

The objective of this trial is to further confirm and assess the efficacy of filiform needle therapy on the common orthopedic pain syndromes and investigate whether or not thumbtack needle therapy could further enhance the clinical efficacy and pain healing effect of the filiform needle therapy.

150 outpatients diagnosed with common orthopedic pain syndromes (Coracoiditis, External humeral epicondylitis, Radial styloid process stenosing tenosynovitis, Flexor tendon stenosing tenosynovitis, Costochondritis and Supraspinal ligament injury) will be recruited. The recruited patient will be divided randomly into (i)Filiform Needle Group (75 cases) and (ii)Filiform Needle supplemented by Thumbtack Intra-dermal Needle Group (75cases) by using computer generated random number.

During the study period, a maximum of two courses of acupuncture therapy, consisting of 7 sessions each, will be administered. Treatment will be given twice per week. After completing the first course of 7 sessions, there will be a break of one week, at the end of which the second course will commence. Treatment will come to a halt as soon as the pain has totally subsided. The aim of treatment is to relieve the pain associated with the common orthopedic syndrome within the shortest period of time.

Questionnaire incorporating The Short-form McGill Pain Form and selected life efficacy questions will be used in this study to quantify the level of pain. Traditional Chinese Medicine(TCM) Syndrome Diagnostic Efficacy Standards and The Guiding Rules of Clinical Research of New Chinese Medicine will be adopted as the standard to observe and evaluate the efficacy of treatment. Patients will be observed and evaluate before and after each treatment and each treatment course. The subjects' level and intensity of pain will be recorded together with the improvement of body mobility and symptoms related to the pain. Follow up will take place 3 months, 6 months and 12 months after treatment completed through phone interview.

Data collected will be analysed by Statistical Product and Service Solutions(SPSS) statistical software, The efficacy of Filiform Needle Therapy and Thumbtack Needle Therapy on Common Orthopedic Pain Syndromes will be objectively assessed and compared.

ELIGIBILITY:
Inclusion Criteria:

* a. Age:>18 years old
* b. Gender: male or female
* c. Duration: not restricted
* d. Comply with Western medicine diagnostic criteria.
* e. Signed the Patient/Subject Consent Form for this study.

Exclusion Criteria:

* a. The disease is not comply with Western diagnostic criteria.
* b. The disease is outside the range of this study.
* c. Acute disease activity phase.
* d. Skin swelling, skin infection, skin active ulcer disease, or local purpura and scar.
* e. Patients with skin allergies, bleeding disorders
* f. Pregnancy, lactating women.
* g. Application of other therapy, the disease has been or is gradually improving.
* h. Chronic wasting disease.
* i. Severe primary diseases of the liver, kidney, hematopoietic system and -endocrine system,
* j. Mental illness.
* k. With other severe diseases, it is difficult to exact evaluate the efficacy and safety of acupuncture.
* l. Not signed the Patient/Subject Consent Form for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change of score on Mcgill pain form (SF) | 1 week
  The change of Score on Mcgill pain form (SF) between baseline and after the 7th treatment will be measured and compared between groups. Should the patient terminate treatment before the 7th treatment, (due to any reason including cure and drop out), the score of the last treatment will be used for analysis.
Change of pain intensity on visual analogue scale (VAS) (1-10) | 1 week
  The change of pain score on VAS scale between baseline and after the 7th treatment will be measured and compared between groups. Should the patient terminate treatment before the 7th treatment, (due to any reason including cure and drop out), the score of the last treatment will be used for analysis. Follow up phone call will be conducted 3 months after the treatment completed for all patients. The VAS score of the treatment position will be recorded to understand the pain remission pattern between groups

SECONDARY OUTCOMES:
The improvement of clinical signs and symptoms | 1 week
  The improvement of clinical signs and symptoms will be compared between groups. The following standard is used to classify improvement of clinical signs and symptoms
  1. Clinically cured: the overall improvement rate of the main symptoms and signs≧95%, normal joint movement.
  2. Significantly improved: the overall improvement rate of the main symptoms and signs≧70%, the joint activities are not limited.
  3. Improved: the overall improvement rate of the main symptoms and signs≧30%, <70%，the Joint activities have been improved.
  4. Inefficacy: the overall improvement rate of the main symptoms and signs <30%, the Joint activities have not been improved.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, Principal Investigator — The University of Hong Kong
Locations (1):
- School of Chinese Medicine, The University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided